CLINICAL TRIAL: NCT00220883
Title: Reproducibility and Inter-Reader Reliability of Electrogastrographic Readings in Normal Subjects and Dyspeptic Patients
Brief Title: Electrogastrogram (EGG) Reproducibility Study: EEG Readings in Normal Subjects and Dyspeptic Patients
Status: Completed | Type: Observational
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Other Study IDs: TU4687
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Electrogastrography

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The primary objective of this study is to determine whether EGG readings obtained from both normal subjects and dyspeptic patients are reproducible from one EGG recording to another on a different day.

The secondary objective of this study is to determine whether the EGG readings are analyzed and diagnosed consistently when reviewed and compared by multiple blinded readers when the same tracing is reviewed.

DETAILED DESCRIPTION:
This is a single-center study. The duration of this trial is estimated to be six months. A total of Forty (40) subjects will be recruited into this study. It will be two Groups; ten (10) normal healthy subjects will be recruited by poster advertisement and thirty (30) patients who either present to the Gastroenterology Department of Temple University Hospital with varying signs, symptoms or complaints of gastric discomfort, or who are scheduled to undergo an EGG test by their Gastroenterologist.

Each study subject/patient will have a total of two (2) EGGs with Water load tests performed for this study. Each EGG exam will be performed approximately one (1) week of each other, but no more than 4 weeks apart, and will be read in a blinded fashion by three (3) separate independent readers, in order to see if the readings are consistent with the previous readings that were obtained, as well as, by the readers themselves (Inter-reader rater reliability). Each reader will be blinded to the subject status (normal/healthy or patient) and also to the specific test they are reading (initial exam [Visit 1], or follow-up exam 1 week after Visit 1 [Visit 2]). All EGG exam results will be coded in order to keep them blind.

ELIGIBILITY:
For normal healthy subjects:

Inclusion Criteria:

1. Male or female patients who are 18 years of age to 72 years of age.
2. Normal healthy subjects with no signs or symptoms of gastrointestinal discomfort.

Exclusion Criteria:

Patients will not be included in this study if they are:

1. < 18 years of age or >72 years of age
2. Subjects with known gastrointestinal or liver cancers, pancreaticobiliary tract diseases, active peptic ulcer disease or uncontrolled lactose intolerance.
3. Subjects with cardiovascular, pulmonary disorders, or subjects with diabetes mellitus, a malignancy or who are known to be HIV positive.
4. Subjects with a history of gastric, intestinal or colonic resections. Subjects who are at less than a three month status for either: post appendectomy, cholecystectomy, or hysterectomy with or without oophorectomy.
5. Subjects who are unable to give informed consent or adequately express their subjective complaints.
6. Subjects who abuse drugs or alcohol.
7. Female subjects who are pregnant.

For functional dyspepsia patients:

Inclusion Criteria:

1. Male or female patients who are 18 to 72 years of age.
2. Patients who present with varying gastric complaints of discomfort
3. Patients who meet all Rome II criteria for functional dyspepsia (see Rome II criteria checklist)

Concomitant medications are allowed during the study period.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-08 (Actual); Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry P Parkman, MD, Principal Investigator — Temple University
Locations (1):
- Temple University School of Medicine, Philadelphia, Pennsylvania, United States